CLINICAL TRIAL: NCT06792240
Title: EVALUATION of IRON INTAKE UPON BLASMA - PHENYLALANINE LEVELS in PHENYLKETONURIA PATIENTS in 3 YEARS LONGITUDINAL RANDOMIZED STUDY
Brief Title: Iron Supplements Effect on B-Phe Levels in PKU Patients During 3 Years Study
Acronym: ISPEK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASST Santi Paolo e Carlo (Other)
Collaborators: Università Luigi Vanvitelli della Campania (Unknown)
Responsible Party: Principal Investigator, Raed Selmi, DR, ASST Santi Paolo e Carlo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43183/2019 - 2019/ST/142
Record Dates: First submitted 2025-01-01; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Phenylketonuria (PKU)
Keywords: PKU; Phe; Iron
MeSH Terms: conditions — Phenylketonurias | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Cohort stydy. The duration of iron supplementation lasted for 3 consecutive months for each patient in Group A. 3 clinical and hematological controls were performed at T0 (the enrolment day), T3 (3 months from T0) and T6 (6 months from T0). This study contains of 84 children (A= 42) Iron Group and (B= 42) control group. As our active protocol at the Metabolic Centre, the patient must do one blood sample / Guthrie card each month to measure only Phe, Tyr levels, and Phe/Tyr Ratio with standardized methods. That allow the researcher to add 4 blood drop samples gathered by Guthrie card (T1, T2, T4, and T5) per each patient during long the study. It is clear now that each participant underwent blood sample collections at T0, T3, and T6 and blood drop sample collections at T1, T2, T4, and T5 using the Guthrie card (TG).
Masking Description: A computer-generated block sequence balanced randomly assigned subjects to two different groups of 42 patients. The investigator who generated the randomization sequence was independent of the research staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group (A) (Experimental): treated with low Phe diet therapy and iron supplementation
  Interventions: Dietary Supplement: iron supplementation
- group (B) (Other): treated only with low Phe diet therapy
  Interventions: Dietary Supplement: control group

INTERVENTIONS:
Dietary Supplement: iron supplementation — The amount of supplementary iron was decided for patients according to the daily requirement (8- 18 mg / day), according to LARN 2012 and (RDAs) for Iron. (25) . This study took in consideration also, the recommendation of the National Institutes of Health iron dietary supplement fact of sheet as reference to calculate iron dose for our candidates because this dose isn't against LARN and more practical to applicate.
  The minimum RDA values is applied, which coincides within the LARN daily requirement limits. (7 mg-18 mg of iron per day). Applying the minimum recommended RDA dose, that can satisfy the daily iron requirement by age, approximating it to be adequate for the clinical dose administered orally once a day (e.g. 1.98 g ==> 2 g, 1.53 g ==> 1.5 g
  Arms: group (A)
Dietary Supplement: control group — Non intervension: Only restricted low and controlled Phe diet therapy
  Arms: group (B)

SUMMARY:
This clinical trial study aims to Evaluate whether iron supplementation for 3 months may help reduce Phe blood concentration in PKU patients by enhancing the hydroxylation of Phe to tyrosine (Tyr).

84 patients affected by PKU with low Phe-controlled diet therapy (aged 3-25 years, both genders, 35 females and 49 males), were randomly enrolled in this 3 years study using Randomized Block Design. Patients were divided in two different groups: group (A) was treated with low Phe diet therapy and iron supplementation while group (B) was treated only with low Phe diet therapy. The duration of iron supplementation was 3 consecutive months for each patient in group (A). During this study, 3 hematological and clinical controls were performed at T0 (the enrolment day), T3 (3 months from T0), and T6 (6 months from T0) another TG was done at T1, T2, T4, and T5. During the clinical control blood samples for phenylalanine, and tyrosine were performed on all patients.

A computer-generated block sequence balanced randomly assigned subjects to two different groups of 42 patients. The investigator who generated the randomization sequence was independent of the research staff. Energy calculation and diet preparation are according to the "Reference intake levels of nutrients and energy for the Italian population (LARN)" and RDA (USA- Recommended Daily Allowance). The patients were informed through the consent form about all study details. The researcher clarified that the iron supplementation was provided to patients for the purpose of studying "Phe" levels, oxidative stress, and inflammatory reactions, and not for treating Anemia before enrolling in this study.

The amount of supplementary iron was decided for patients according to the daily requirement (8- 18 mg / day), according to LARN 2012 and (RDAs) for Iron.

The number of patients in group A (42 patients) that consumed iron of 1 sac (14 mg/day) was 26 patients (61.9 %), of them 18 males and 8 females, in comparison with patients that consumption 1 sac an alternative day (14mg/every 2 days) = (7 mg/day- ½ sac/ day) was 16 patients (38.1%) of them 9 males and 7 females.

Conclusions and Relevance:

* Our data suggests that regular iron supplementation could be needed to obtain better metabolic control in PKU patients, as it seems to be directly linked to lowering blood Phe levels. Thus, support that iron supplementation to PKU patients plays a relevant role for accurate function of PAH enzyme, probably represents one activator and it may can help to decrease the b-Phe value near to the normal range with - 46.7% of Phe, - 74.52% of Phe/Tyr ratio and increase 91.07% Tyr all with (P<00.1) from the basal values
* It is also confirmed that oral iron supplementation with FERALGINE (FB + SA) to these patients could represent "as part of a comprehensive PKU management strategy" considering the high effectiveness and tolerability profile.
* additional study is required before the information should be used support our results The investigators declare that no conflict of interest.

DETAILED DESCRIPTION:
Introduction: Phenylketonuria (PKU) (OMIM 261600) is an autosomal recessive congenital metabolic disease with an average of about 1:10,000 newborns, characterized by Phe accumulation in the body due to deficiency of the PAH, Most cases (98%) of PKU/HPA result from mutations in the phenylalanine hydroxylase (PAH) gene which locates on the chromosom e 12q24.1, that lead to deficient or absent activity PAH enzyme (EC 1.14.16.1). The remaining cases (2%) arise due to a block in the metabolism of Tetrahydrobiopterin (BH4) the PAH cofactor. Normal blood levels of Phe are <120 mmol/L, Based on blood Phe concentrations, PAH deﬁciency can be classiﬁed into classic PKU (Phe >1200 μmol/L), mild PKU (Phe = 600-1200 μmol/L) and mild Hyperphenylalaninemia (MHP) (Phe = 120 - <600 μmol/L). High concentration of Phe in blood (>360 μmol/L) at neonatal age, could lead to irreversible brain damage, but it can be prevented by early diagnosis, thanks to newborn screening and initiation of Phe-restricted diets.

The main source of natural nutrients, especially Iron (Fe), Vitamin B12 (vit B12), and Vitamin D (vit D) in normal children's diet are foods containing proteins; so, its restriction in the dietary management of PKU can lead to essential element's deficiency, anaemia, irreversible neurological defects and failure to thrive. Nowadays, these elements can be supplemented through special diet therapy. Diagnosis of HPA is made based on an elevated blood Phe concentration on a repeat blood sample confirmed genetically. The upper reference limit for Phe in whole blood or plasma in neonates is 120 μmol/L(9). All patients, at newborn screening, with plasma Phe levels, of more than 360 μmol/L, must initiate restricted low and controlled Phe diet therapy (RLCPDT) as early as possible to prevent above mentioned complications. The dietary scheme includes also other supplementations of Docosahexaenoic acid (DHA), vitamins, and other nutrients. Fe is not yet considered a recommended supplementation to PKU patients although most of our patients are supplanted with this micronutrient due to the finding of anaemia. the investigators noted that the patients supplanted with iron have consequentially reduced Phe plasma levels. This may be conceded with the fact that the investigators realized this study to confirm the relation of Iron supplementation with P-Phe levels.

The PAH enzyme is tetrameric and contains three major domains including a regulatory, a small tetramerization and a catalytic domain that contains the active site that includes a ferrous iron (Fe) prosthetic group bound to three charged aminoacid residues. So that PAH enzyme performs its hydroxylation function correctly, it requires the presence of iron, oxygen, and a cofactor, Tetrahydrobiopterin (BH4) to hydroxylase Phe in Tyr.

Based on these structural and functional considerations, it is hypothesized that iron supplementation in PKU patients can enhance the activity of the PAH enzyme, consequently reducing their blood levels of Phe. At the researcher's consciousness this study is the first to be applied to PKU human patients.

Lectures studies regarding iron and PKU: J. L. Bodley, revealed a high incidence of low stores of iron in 53 low-phenylalanine diet PKU patients in a retrospective study. These findings suggest that the current dietary management of PKU is associated with an increased risk for low iron store depletion.

Mackler et al, analyzed a pre-clinical observation study evidenced that, the concentrations of plasma phenylalanine (P-Phe) were markedly elevated in iron-deficient rats and appeared to vary directly with the degree of iron deficiency. Plasma concentrations of Phe returned to control levels within one week after treatment of the iron-deficient rats with iron. The elevated levels of P-Phe were probably not produced by a deficiency in liver PAH because levels of activity of the enzyme were found to be normal in the livers of analyzed animals.

Gropper SS et al, demonstrated that, the P-Phe concentrations are associated with hepatic iron content in a murine model for phenylketonuria.

Ferrous Bisglycinate (FB) and Sodium Alginate (SA) combination is The first choice as iron supplementation: The researcher did keen research on the various types of iron supplementations available in commerce. After deep analysis was conducted the Iron amino acid chelates, as Iron Glycinate Chelates (IGC) group, are developed to be used as food fortificants and therapeutic agents in the prevention and treatment of iron deficiency anemia. The absorption of iron from Ferrous Bisglycinate (FB) is regulated through the same physiological mechanisms as other inorganic forms of iron. Following oral administration, FB contributes to the intestinal intraluminal pool of inorganic non-heme iron and is absorbed intact into the mucosal cells of the intestine. Subsequently, it is hydrolyzed into its iron and glycine components. Its safety and maximum tolerable intake have been reviewed and evaluated by several scientific committees.

The important factor that helps us to choose FB is that it has been used in the fortification of foods providing between 2 and 23 mg/day of supplemental dietary iron without any reports of adverse effects. Furthermore, FB has been well-tolerated as a dietary iron supplement, providing approximately 15 to 120 mg of iron per day, across various population groups, including adult males, pregnant females, non-pregnant females with normal iron levels, and particularly among iron-deficient young children.

The stability of FB (by the addition of the product to milk, yogurt, corn flour, and margarine) and the lack of potential for interaction of FB with these foods (lipid peroxidation) have been tested at various times/temperatures. There is no evidence to indicate the occurrence of reactions of FB with components of these foods, and it is confirmed that FB provides a highly bio-available and stable source of iron.

FB is protected from interaction with dietary inhibitors of iron absorption such as Phytate and the iron absorption from this molecule is normally down-regulated as iron stores increase.

The combination of (FB + SA) oral supplementation formula has been demonstrated to be more bioavailable, safer and tasteful when compared to FB alone. Since (FB + SA) are present in 1 to 1 ratio, every little particle of the powder has the same morphology and quantity of the two different co-processed substances. The new "co-processed compound", obtained by spray drying technology, confers to the iron powder an increase and uniform superficial area and, consequently, quick and more extensive iron absorption together with an increased gastrointestinal protection. In the same time, the uniform presence of SA in this product, allows the FBC to be released more constantly and slowly when confronted to FB alone and let the Divalent Metal Transporter 1 (DMT-) receptors to better uptake iron. DMT1 receptor saturation could be a limit in oral iron bioavailability that could be exceeded by FERALGINE (FB + SA). In fact, slowly availability of iron by FB+ SA administration could result in DMT-1 unsaturation with the consequence of increasing iron bioavailability.

Iron Bisglycinate product analysis: Considering our previous clinical experiences with FB alone in the previous years and our experiences with the new compound containing a spray-drying technology co-processed substance (FB + SA named Feralgine) in a 1 to 1 ratio supporting more bioavailability and less gastrointestinal adverse events for this research the investigators decided to use only FERALGINE effervescent sachets.

Our clinical experience was also supported by the published literature. The researcher decided to exclude oral capsule and tablet forms because children have difficulty swallowing these preparations and exclude oral drops because it is not adapted to teenagers and adult patients resulting in low domiciliary compliance, especially for long-term use, Considering that the formulation of effervescent sachets containing Feralgine (FB + SA), a compound more bioavailable, with high gastrointestinal tolerability, more tasteful, and able to increase domiciliary compliance especially for long-term use, the investigators decided to use only available Feralgine preparation containing effervescent sachets with 14 mg of elemental iron according to patient's age and weight.

Patients and Methods:

* Study population The study was performed as a 3 years longitudinal interventional randomized parallel assignment clinical trial involving 84 PKU patients in diet therapy with low and controlled Phe intake divided into two groups, 42 patients (group A) with iron supplementation in comparison with other 42 patients (group B) without iron supplementation.
* Sample size and randomization The sample size was calculated regards the duration of the study, availability, heterogeneity of patients, and our resources. To detect a 20% or greater change in mean plasma Phe levels at the end of the intervention period in the iron-supplemented group compared to the control group. For these 84 children (42 per group) were recruited.

A computer-generated block sequence balanced randomly assigned subjects to two different groups of 42 patients for each. An independent investigator-generated the randomization sequence separate from the researcher. https://www.sealedenvelope.com was used for the generation of the randomization lists. Children were assigned to the intervention group (A) or to the control group (B) through lists stratified by sex and age (3-6, 7-10, 11-14, 15-25 years), in blocks of 4 units.

The setting of participants: The study was approved by the Italian Ethics Committee (ASST-SANTI PAOLOCARLO), Protocol No: 43183/2019 in date 10/10/2019 -and all participants or their legal representative approved and signed the informed written consent on enrolment day. All participants in the study satisfied eligibility for the study.

All experimental procedures adhered to the Declaration of Helsinki and all assessments were performed by trained medical staff. The present study has been examined PKU patients who were aged from 3 to 25 years, diagnosed and followed by the ASST Santi Paolo and Carlo, Pediatrics department of San Paolo Hospital at Milan the Lombardy Regional Centre.

The duration of iron supplementation lasted for 3 consecutive months for each patient in Group A. 3 clinical and hematological controls were performed at T0 (the enrolment day), T3 (3 months from T0) and T6 (6 months from T0). This study contains of 84 child (A= 42) Iron Group and (B= 42) control group. As our active protocol at Metabolic centre, the patient must do one blood sample / Guthrie card each month to measure only Phe, Tyr levels and Phe/Tyr Ratio with standardized methods. That allow the researcher to add 4 blood drop samples gathered by Guthrie card (T1, T2, T4 and T5) per each patient during long the study. It is clear now that each participant underwent to blood sample collections at T0, T3, and T6 and blood drop sample collections at T1, T2, T4, and T5 using the Guthrie card (TG). A computer-generated block sequence balanced randomly assigned subjects to two different groups of 42 patients. The investigator who generated the randomization sequence was independent of the research staff. Energy calculation and diet preparation are according to the "Reference intake levels of nutrients and energy for the Italian population (LARN)" and RDA (USA- Recommended Daily Allowance). The patients were informed through the consent form about all study details. The researcher clarified that the iron supplementation was provided to patients for the purpose of studying "Phe" levels, oxidative stress, and inflammatory reactions, and not for treating Anemia before enrolling in this study.

Normal values of blood analysis (ASST-Santi Paolo and Carlo - Milan): Phenylalanine Phe Umol/L (n.v < 120), Tyrosine Tyr Umol/L (n.v 30-120) , PHE/TYR Ratio (n.v <0.9) Intervention and supplements: The amount of supplementary iron was decided for patients according to the daily requirement (8- 18 mg / day), according to LARN 2012 and (RDAs) for Iron . This study took in consideration also, the recommendation of the National Institutes of Health iron dietary supplement fact of sheet as reference to calculate iron dose for our candidates because this dose isn't against LARN and more practical to applicate.

The minimum RDA values is applied, which coincides within the LARN daily requirement limits. (7 mg-18 mg of iron per day). Applying the minimum recommended RDA dose, that can satisfy the daily iron requirement by age, approximating it to be adequate for the clinical dose administered orally once a day (e.g. 1.98 g ==> 2 g, 1.53 g ==> 1.5 g). Taking into consideration the iron supplemented in the low Phe dietary therapy, so as not to exceed the maximum daily dose required by age and sex according to LARN and RDA.

Patients whose enrolled in the group supplemented with iron (group A) was provided free of charge with the total 3 months doses. The Iron cost tolerated by the researcher. The supplement's trade name was kept anonymous to prevent conflicts of interest and avoid any form of advertising.

The number of patients in group A (42 patients) that consumed iron of 1 sac (14 mg/day) was 26 patients (61.9 %), of them 18 males and 8 females, in comparison with patients that consumption 1 sac an alternative day (14mg/every 2 days) = (7 mg/day- ½ sac/ day) was 16 patients (38.1%) of them 9 males and 7 females.

Statistical analyses: Descriptive data was reported as mean (standard deviation [SD], median (interquartile range [IQR] 25th-75th percentile) or number of observations and percentage. Shapiro Wilk Test was used to assess distribution. Longitudinal changes in Phe and oxidative stress parameters, within group, Inter and Intra subject Variability were tested using Student's t-test for paired data and the Wilcoxon test, when appropriate. Univariate comparisons between the intervention and control groups were performed: for continuous variables by unpaired Student's t-test or Mann-Whitney test and/or analysis of variance for repeated measures; to evaluate the differences between two groups for continuous variables the investigators used the Mann Whitney test, ANOVA repeated measure when appropriate. Multiple binary logistic regression analyses were performed to evaluate the dependence of an independent variables on a dependent variables. Friedman Test model is adjusted for confounding factors, were used to evaluate the effect of iron supplementation on plasma Phe levels and to estimate the corresponding odds ratio (OR ) and its 95% confidence interval. A statistical significance level is p ≤ 0.05 (two-tailed test) was considered. Statistical analyzes was performed with SPSS, version 25.0 (SPSS Inc, Chicago, IL) for Windows (Microsoft Corporation, Redmond, WA).

ELIGIBILITY:
Inclusion Criteria:

* • The diagnosis of PKU must be made before 28 days of life, and confirmed genetically,

  * At the diagnosis, patients' plasma Phe levels have at least two values ≥ 360 µmol/l.
  * Phe low diet therapy started immediately after diagnosis confirmation.
  * The age of participants, male or female, between 3-25 years old at scheduled Day one.
  * Participants have no other diseases,
  * Mean Phe levels should be between 120-360 µmol/l, within 3 months, before the Day 1.

Exclusion Criteria:

* • Diagnosed by any type of anemia, hematological, chronic or gastrointestinal diseases.

  * If acute infection has been diagnosed the Day 1.
  * Administration iron less than 3 months before the start the study.
  * Known hypersensitivity to other approved formulations of Ferrous Bisglycinate.
  * Current use of experimental or unregistered drugs that may affect the study outcomes.
  * Inability to comply with study procedures or inability to tolerate oral intake.
  * History of organ transplantation.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
a significant decrease of Plasma Phe levels in Group A | The duration of iron supplementation lasted for 3 consecutive months for each patient in Group A. 3 clinical and hematological controls were performed at T0 (the enrolment day), T3 (3 months from T0) and T6 (6 months from T0).
  The outcome evidenced using Chi-square of di Pearson test a significant decrease (p<0.001) - 46.7% of Phe, - 74.52% of Phe/Tyr ratio (population supplemented with Iron shows a significant metabolic improvement; in particular, Phe values. Used SPSS software and Prism software.

CONTACTS AND LOCATIONS:
Overall Officials: Raed Selmi, MD-PhD, Principal Investigator — ASST Santi Paolo e Carlo
Locations (1):
- ASST-Santi Paolo e Carlo, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Results will be published by the investigators in academic journals.

REFERENCES:
- [Background] Institute of Medicine. Food and Nutrition Board. Dietary Reference Intakes for Vitamin A, Vitamin K, Arsenic, Boron, Chromium, Copper, Iodine, Iron, Manganese, Molybdenum, Nickel, Silicon, Vanadium, and Zinc : a Report of the Panel on Micronutrients external link disclaimer. Washington, DC: National Academy Press; 2001
- [Background] Chace DH, Hannon WH. Filter Paper as a Blood Sample Collection Device for Newborn Screening. Clin Chem. 2016 Mar;62(3):423-5. doi: 10.1373/clinchem.2015.252007. Epub 2016 Jan 21. No abstract available. PMID 26797689
- [Background] Gervasi GB, Baldacci M, Bertini M. Feralgine® a new co-processed substance to improve oral iron bioavailability, taste and tolerability in iron deficiency patients. Arch Med. 2016;8:13-16. 25) LARN Livelli di Assunzione di Riferimento di Nutrienti ed energia per la popolazione Italiana ( https://sinu.it/tabelle-larn-2014/)
- [Background] Baldacci M, Gervasi GB, Bertini M. Iron deficiency anemia (ida) and iron deficiency (id): are alginates a good choise to improve oral iron bioavailability and safety? J TranslSci. 2018;4:1-3. DOI: 10.15761/JTS.1000210
- [Background] Allen LH. Advantages and limitations of iron amino acid chelates as iron fortificants. Nutr Rev. 2002 Jul;60(7 Pt 2):S18-21; discussion S45. doi: 10.1301/002966402320285047. No abstract available. PMID 12141594
- [Background] Soldin OP, Bierbower LH, Choi JJ, Choi JJ, Thompson-Hoffman S, Soldin SJ. Serum iron, ferritin, transferrin, total iron binding capacity, hs-CRP, LDL cholesterol and magnesium in children; new reference intervals using the Dade Dimension Clinical Chemistry System. Clin Chim Acta. 2004 Apr;342(1-2):211-7. doi: 10.1016/j.cccn.2004.01.002. PMID 15026283
- [Background] Bovell-Benjamin et al., 2000; Layrisse et al., 2000; García-Casal and Layrisse, 2001; Jeppsen, 2001
- [Background] Opinion of the Scientific Panel on Food Additives, Flavourings, Processing Aids and materials in Contact with Food on a request from the Commission related to Ferrous bisglycinate as a source of iron for use in the manufacturing of foods and in food supplements. Question number EFSA-Q-2005-039 . Adopted on 6 January 2006 by written procedure. https://efsa.onlinelibrary.wiley.com/doi/epdf/10.2903/j.efsa.2006.299
- [Background] Vargas CR, Wajner M, Sitta A. Oxidative stress in phenylketonuric patients. Mol Genet Metab. 2011;104 Suppl:S97-9. doi: 10.1016/j.ymgme.2011.07.010. Epub 2011 Jul 22. PMID 21813309
- [Background] Guerra IMS, Ferreira HB, Neves B, Melo T, Diogo LM, Domingues MR, Moreira ASP. Lipids and phenylketonuria: Current evidences pointed the need for lipidomics studies. Arch Biochem Biophys. 2020 Jul 30;688:108431. doi: 10.1016/j.abb.2020.108431. Epub 2020 May 24. PMID 32461102
- [Background] Gropper SS, Yannicelli S, White BD, Medeiros DM. Plasma phenylalanine concentrations are associated with hepatic iron content in a murine model for phenylketonuria. Mol Genet Metab. 2004 May;82(1):76-82. doi: 10.1016/j.ymgme.2004.01.017. PMID 15110326
- [Background] Mackler B, Person R, Miller LR, Finch CA. Iron deficiency in the rat: effects on phenylalanine metabolism. Pediatr Res. 1979 Sep;13(9):1010-1. doi: 10.1203/00006450-197909000-00012. PMID 503651
- [Background] Bodley JL, Austin VJ, Hanley WB, Clarke JT, Zlotkin S. Low iron stores in infants and children with treated phenylketonuria: a population at risk for iron-deficiency anaemia and associated cognitive deficits. Eur J Pediatr. 1993 Feb;152(2):140-3. doi: 10.1007/BF02072491. PMID 8444222
- [Background] Robin A Williams, et al (Scriver CR, Kaufman S. Hyperphenylalaninemia: phenylalanine hydroxylase deficiency. In: Scriver CR, Beaudet AL, Sly WS, Valle D, Childs B, Kinzler K, Phenylketonuria: An Inborn Error of Phenylalanine Metabolism. Vogelstein B, editors. The Metabolic and Molecular Bases of Inherited Disease. 8th ed. New York: McGraw- Hill; 2001. p. 1667-724).
- [Background] Navarro G, Gomez-Autet M, Morales P, Rebassa JB, Llinas Del Torrent C, Jagerovic N, Pardo L, Franco R. Homodimerization of CB2 cannabinoid receptor triggered by a bivalent ligand enhances cellular signaling. Pharmacol Res. 2024 Oct;208:107363. doi: 10.1016/j.phrs.2024.107363. Epub 2024 Aug 22. PMID 39179054
- [Background] Knox WE. Retrospective study of phenylketonuria: relation of phenylpyruvate excretion to plasma phenylalanine. PKU newsletter 1970;2
- [Background] Hanley WB, Linsao L, Davidson W, Moes CA. Malnutrition with early treatment of phenylketonuria. Pediatr Res. 1970 Jul;4(4):318-27. doi: 10.1203/00006450-197007000-00002. No abstract available. PMID 5447890
- [Background] Lichter-Konecki U, Vockley J. Phenylketonuria: Current Treatments and Future Developments. Drugs. 2019 Apr;79(5):495-500. doi: 10.1007/s40265-019-01079-z. PMID 30864096
- [Background] Blau N, et al. Disorders of phenylalanine and tetrahydrobiopterin metabolism. In: Blau N, Hoffmann GF, Leonard J, Clarke JTR, editors. Physician's guide to the treatment and follow-up of metabolic diseases. Berlin: Springer; 2006. p. 25-34
- [Background] Fitzpatrick PF. Mechanism of aromatic amino acid hydroxylation. Biochemistry. 2003 Dec 9;42(48):14083-91. doi: 10.1021/bi035656u. No abstract available. PMID 14640675
- [Background] Nenad Blau. Phenylketonuria and BH4 deficiencies- UNI-MED 2010. ISBN: 978-1-84815-162-8
- [Background] Matthew M. Phenylketonuria: Defects in Amino Acid Metabolism. South Carolina Journal of Molecular Medicine (SCJMM) 5:57-61; 2004
- [Background] Williams RA, Mamotte CD, Burnett JR. Phenylketonuria: an inborn error of phenylalanine metabolism. Clin Biochem Rev. 2008 Feb;29(1):31-41. PMID 18566668
- See also: Reference range of ferritin — https://emedicine.medscape.com/article/2085704-overview